CLINICAL TRIAL: NCT05214508
Title: Serum Interleukin 6 in Chronic Obstructive Pulmonary Disease Patients and Its Relation to Severity and Acute Exacerbation
Brief Title: Serum Interleukin 6 in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Fatma Gamal Mohamed, assisstant lecturer, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: faculty of medicine
Record Dates: First submitted 2022-01-14; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Chronic Obstr Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD patient (Active Comparator): COPD patients diagnosed based on spirometry, PFT and history
  Interventions: Diagnostic Test: interleukin 6
- Control (No Intervention): Healthy volunteers

INTERVENTIONS:
Diagnostic Test: interleukin 6 — assessment of serum IL-6 by ELISA
  Arms: COPD patient

SUMMARY:
The aim of this study is to estimate level of IL 6 in COPD patients and its relation to COPD severity and acute exacerbation.

DETAILED DESCRIPTION:
1. A detailed clinical history was be carried out for every patient. In the clinical history, duration of COPD with a history of exacerbation and treatment will be elicited. History of the presence of risk factors such as smoking, exposure to fumes (biomass), and the presence of any other chronic disease were be inquired.
2. Thereafter, the detailed physical examination also had been carried out.
3. Pulmonary function test was performed by master screen NO : 781040 (care fusion) Measurements were obtained for FVC,FEV1,Ratio between them, PEF,FEF25%,FEF50% ,and FEF75% (The readings for FEV1 and Ratio were the ones included in the statistical analysis as indices for obstructive pattern of respiration).
4. Labs including Complete blood count, urea, and serum creatinine ,ESR was done for all patients
5. Exercise capacity by six minutes' walk test.
6. Dyspnea score by MMRC score.
7. Health state assessment by CAT score

3- 8- Determination of IL 6 serum levels. by sandwich enzyme-linked immunosorbent assay (ELISA). The detection range (0.2 ng/L- 8ng/L)

ELIGIBILITY:
Inclusion Criteria:

1. All patients aged >40 years and <80 years, of both gender
2. Diagnosed to have COPD according to GOLD 2019 by spirometry
3. Given the consent for participation in the study

Exclusion Criteria:

1- Any patient with systemic inflammation as

1. Bronchial asthma,
2. rheumatoid arthritis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
measure level of IL-6 | 9 monthes
  using ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Laila Anwar Sharawy, Study Director — Beni Suef faculty of medicine
Locations (1):
- Beni Suef university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Available for all researchers
Supporting Information: Study Protocol, SAP
Time Frame: 3/2022 for 2 years
Access Criteria: All